CLINICAL TRIAL: NCT00820846
Title: A Phase 2a Clinical Trial to Evaluate the Safety and Immunogenicity of a Prime-boost Vaccine Regimen of pGA2/JS7 DNA and MVA/HIV62, in Healthy, HIV Uninfected Vaccinia-naive Adult Participants
Brief Title: Safety of and Immune Response to a Prime-Boost Vaccine Regimen in HIV-Uninfected Vaccine-Naive Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 205; 10658 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part A, Group 1 (Experimental): Participants will receive two injections of the pGA2/JS7 DNA vaccine and then two injections of the MVA/HIV62 vaccine
  Interventions: Biological: pGA2/JS7 DNA vaccine; Biological: MVA/HIV62 vaccine
- Part A, Group 2 (Placebo Comparator): Participants will receive four placebo injections
  Interventions: Biological: Placebo
- Part B, Group 3 (Experimental): Participants will receive two injections of the pGA2/JS7 DNA vaccine and then two injections of the MVA/HIV62 vaccine
  Interventions: Biological: pGA2/JS7 DNA vaccine; Biological: MVA/HIV62 vaccine
- Part B, Group 4 (Experimental): Participants will receive three injections of the MVA/HIV62 vaccine and one injection of the placebo
  Interventions: Biological: Placebo; Biological: MVA/HIV62 vaccine
- Part B, Group 5 (Placebo Comparator): Participants will receive four placebo injections
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: pGA2/JS7 DNA vaccine — 1 mL of pGA2/JS7 DNA vaccine
  Arms: Part A, Group 1; Part B, Group 3
Biological: Placebo — 1 mL of sodium chloride for injection
  Arms: Part A, Group 2; Part B, Group 4; Part B, Group 5
Biological: MVA/HIV62 vaccine — 1 mL of recombinant modified vaccinia Ankara/HIV clade B gag-pol-env (MVA/HIV62)
  Arms: Part A, Group 1; Part B, Group 3; Part B, Group 4

SUMMARY:
The purpose of this study is to evaluate the safety of and immune response to a two-vaccine regimen in healthy, HIV-uninfected adults who have never received an HIV preventive vaccine before.

DETAILED DESCRIPTION:
Some of the first HIV vaccines were designed to trigger neutralizing antibody responses as a way to prevent HIV infection. Unfortunately, the first versions of these vaccines were not able to achieve their desired response. An alternative strategy to the antibody approach is the stimulation of HIV-specific CD8 T-lymphocyte (CTL) responses. CTL responses were previously demonstrated to play an important role in the control of simian immunodeficiency virus (SIV), the HIV equivalent seen in rhesus macaque monkeys. Additionally, other studies suggest CTLs play an important role in viral control during chronic infection. Based on this information, several groups have shifted their focus to the development of CTL-based vaccines, some of which have entered advanced clinical trials.

A DNA/rMVA vaccine strategy is structured to bring about both T-cell and antibody responses. The primary vaccination is DNA based and will express only HIV proteins as a way to produce an HIV-focused immune response. An rMVA vaccine strategy expresses both HIV and MVA proteins and may amplify the focused response of a DNA vaccination. Participants in this study will receive either a combined DNA/rMVA vaccine strategy, in which they receive both types of vaccines; an rMVA vaccine strategy, in which they receive only the rMVA vaccine; or a placebo. The DNA and rMVA are physically two different vaccinations given at separate times, but in the DNA/rMVA group, they will be used together to make up one preventive regimen. Both vaccine components express noninfectious virus-like particles.

This study is a multicenter, randomized study that is conducted in two parts and comprised of five groups. In all groups, participants will receive four injections. In Part A, Groups 1 and 2 will be compared. In Group 1, participants will receive two shots of the DNA vaccine and two shots of the rMVA vaccine. In Group 2, participants will receive four placebo injections. In Part B, Groups 3, 4, and 5 will be compared. In Group 3, the combination vaccine strategy will be used again; in Group 4, a single-vaccine strategy of three injections of the rMVA vaccine and one injection of placebo will be given; and in Group 5, participants will again receive four placebo injections. The study will last for a total of 12 months for participants, including enrollment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research center and willing to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: completion of a questionnaire prior to first vaccination; demonstration of understanding for all questionnaire items answered incorrectly
* Willingness to receive HIV test results
* Good general health as shown by medical history, physical exam, and screening laboratory tests
* Certain specified laboratory values. More information on this criterion can be found in the study protocol.
* If pregnancy is possible, must agree to use contraception from at least 21 days prior to enrollment through the last protocol visit for sexual activity that could lead to pregnancy. More information on this criterion can be found in the study protocol.
* Willingness to discuss HIV infection risks, amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit, and willing to continue annual follow-up contact after the last required protocol clinic visit for a total of 5 years following enrollment
* Assessed by clinic staff as being at "low risk" of HIV infection on the basis of sexual behaviors within the 12 months prior to enrollment. More information on this criterion can be found in the study protocol.

Exclusion Criteria:

* HIV vaccine(s) or other experimental vaccines, received in a prior HIV vaccine trial. More information on this criterion can be found in the study protocol.
* Receipt of smallpox vaccination
* Excessive alcohol use, frequent binge drinking, chronic marijuana abuse, or use of any other illicit drugs, such as cocaine or methamphetamine, within the past 12 months
* History of newly acquired or newly diagnosed syphilis; history of newly acquired gonorrhea, nongonococcal urethritis, herpes simplex virus type 2 (HSV2), chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis,epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B within the past 12 months
* Immunosuppressive medication received within 168 days before first vaccination. Certain medications are excluded from this criterion; more information can be found in the study protocol.
* Blood products received within 120 days before first vaccination
* Immunoglobulin received within 60 days before first vaccination
* Live attenuated vaccines other than influenza vaccine received within 30 days before first vaccination or scheduled within 14 days after injection
* Influenza vaccine or any vaccines that are not live attenuated and were received within 14 days prior to first vaccination or that are scheduled within 14 days after injection
* Allergy treatment with antigen injections within 30 days before first vaccination or scheduled within 14 days after injection
* Intent to participate in another study of an investigational research agent during the planned duration of this study
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Clinically significant medical condition. More information on this criterion can be found in the study protocol.
* Any medical, psychiatric, or social condition or occupational or other responsibility that in the opinion of the investigator might interfere with the study protocol
* Serious adverse reactions to vaccines. More information on this criterion can be found in the study protocol.
* Allergy to eggs and/or egg products
* History of or known active cardiac disease. More information on this criterion can be found in the study protocol.
* Participants who have two or more of the following cardiac risk factors: (1) participant report of history of elevated blood cholesterol defined as fasting low-density lipoprotein (LDL) greater than 160 mg/dL; (2) first degree relative (e.g., mother, father, sister, or brother) who had coronary artery disease before the age of 50 years; (3) current smoker; or (4) body mass index greater than or equal to 35.
* Electrocardiogram (ECG) with clinically significant findings. More information on this criterion can be found in the study protocol.
* Autoimmune disease
* Immunodeficiency
* Asthma other than mild, well-controlled asthma. More information on this criterion can be found in the study protocol.
* Diabetes mellitus, type 1 or type 2, including cases controlled with diet alone. Those with a history of isolated gestational diabetes are not excluded.
* Thyroidectomy or thyroid disease requiring medication during the last 12 months
* Angioedema within the last 3 years if episodes are considered serious or have required medication within the last 2 years
* Hypertension. More information on this criterion can be found in the study protocol.
* Body mass index greater than or equal to 40
* Bleeding disorder diagnosed by a doctor
* Malignancy. Participants with surgical excisions and subsequent observation periods, that in the investigator's estimation have a reasonable assurance of sustained cure or are unlikely to recur during the period of study, are not excluded.
* Seizure disorder, unless the participant has not required medication or had a seizure within the last 3 years.
* Asplenia
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 299 (Actual)
Dates: Start 2009-01; Primary Completion 2012-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Frequency of severe local and systemic reactogenicity signs and symptoms | Throughout study
Frequency of adverse events and assessed relationship to study products | Throughout study
Laboratory measures of safety, including boxplots of white blood cells (WBC), neutrophils, lymphocytes, hemoglobin, platelets, alanine aminotransferase (ALT), creatinine, and cardiac troponin results at baseline and following vaccination | At study entry and following vaccinations
Number of participants with early discontinuation of vaccinations, by treatment group and reason for discontinuation | Throughout study

SECONDARY OUTCOMES:
Responses to individual HIV potential T-cell epitope (PTE) peptide pools representing Env, Gag, and Pol | Throughout study
Percentage of responding CD4+ and CD8+ T cells producing interferon (IFN)-gamma, interleukin (IL)-2, tumor necrosis factor (TNF)-alpha, CD57, perforin, or granzyme B or demonstrating other functions | Measured at study completion
Frequency and titer of humoral responses detected by HIV binding antibody assays to p55 Gag and gp140 Env | Measured at study completion
Frequency of vaccine-induced positive results with end of study HIV serological testing by commercial assays | Measured at study completion
Frequency of CD4+ T-cell responses | Measured 2 weeks following last MVA vaccination
Frequency of CD8+ T-cell responses | Measured 2 weeks following last MVA vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Goepfert, MD, Study Chair — UAB, Div. of Infectious Diseases
Locations (12):
- United States (10):
  - Alabama CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington
- Peru (2):
  - ACSA CRS, Iquitos, Maynas
  - Barranco CRS, Lima

REFERENCES:
- [Background] Miedema F. A brief history of HIV vaccine research: stepping back to the drawing board? AIDS. 2008 Sep 12;22(14):1699-703. doi: 10.1097/QAD.0b013e3283021a61. PMID 18753857
- [Background] Rerks-Ngarm S, Brown AE, Khamboonruang C, Thongcharoen P, Kunasol P. HIV/AIDS preventive vaccine 'prime-boost' phase III trial: foundations and initial lessons learned from Thailand. AIDS. 2006 Jul 13;20(11):1471-9. doi: 10.1097/01.aids.0000237362.26370.f8. No abstract available. PMID 16847401
- [Background] Goepfert PA, Elizaga ML, Seaton K, Tomaras GD, Montefiori DC, Sato A, Hural J, DeRosa SC, Kalams SA, McElrath MJ, Keefer MC, Baden LR, Lama JR, Sanchez J, Mulligan MJ, Buchbinder SP, Hammer SM, Koblin BA, Pensiero M, Butler C, Moss B, Robinson HL; HVTN 205 Study Group; National Institutes of Allergy and Infectious Diseases HIV Vaccines Trials Network. Specificity and 6-month durability of immune responses induced by DNA and recombinant modified vaccinia Ankara vaccines expressing HIV-1 virus-like particles. J Infect Dis. 2014 Jul 1;210(1):99-110. doi: 10.1093/infdis/jiu003. Epub 2014 Jan 7. PMID 24403557
- [Derived] Huang Y, Zhang L, Janes H, Frahm N, Isaacs A, Kim JH, Montefiori D, McElrath MJ, Tomaras GD, Gilbert PB. Predictors of durable immune responses six months after the last vaccination in preventive HIV vaccine trials. Vaccine. 2017 Feb 22;35(8):1184-1193. doi: 10.1016/j.vaccine.2016.09.053. Epub 2017 Jan 25. PMID 28131393